CLINICAL TRIAL: NCT00014105
Title: Phase I/II Trial of Temozolomide and Carboplatin in Recurrent Glioblastoma Multiforme
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atlantic Health System (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068432; NYU-9948; SPRI-NYU-9948; NCI-G00-1907; NCI-V01-1650
Record Dates: First submitted 2001-04-10; First posted 2004-02-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2002-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carboplatin; Temozolomide

INTERVENTIONS:
Drug: carboplatin
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy in treating patients who have recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of temozolomide and carboplatin in patients with recurrent glioblastoma multiforme. II. Determine the acute and long-term toxic effects of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine the potential of either a pharmacokinetic- or pharmacodynamic-mediated drug interaction in patients treated with this regimen. V. Determine the objective response rate in patients treated with the established MTD of this regimen. VI. Determine time to tumor progression and survival in patients treated with this regimen.

OUTLINE: This is a dose-escalation study. Patients are stratified according to prior nitrosourea-based chemotherapy (yes vs no). Patients receive carboplatin IV over 30 minutes on day 1 and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients with a persistent response may continue to receive temozolomide only for an additional 6 courses. Cohorts of 3-6 patients receive escalating doses of carboplatin and temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive carboplatin and temozolomide at the recommended phase II dose.

PROJECTED ACCRUAL: A total of 13-70 patients (3-30 for phase I and 10-40 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent glioblastoma multiforme Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 70-100% Life expectancy: At least 15 weeks Hematopoietic: Granulocyte count greater than 1,500/mm3 Hemoglobin at least 10.0 g/dL Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No myocardial infarction within the past 6 months No congestive heart failure requiring therapy Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No active or uncontrolled infection No psychiatric disorders that would preclude study No other severe concurrent disease that would preclude study No frequent vomiting or other medical condition that would interfere with oral medication administration (e.g., partial bowel obstruction) No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent sargramostim (GM-CSF) Chemotherapy: No prior temozolomide No prior platinum-based chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Recovered from prior major surgery Other: Recovered from prior therapy No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Gruber, MD, Study Chair — NYU Langone Health
Locations (1):
- Overlook Hospital, Summit, New Jersey, United States